CLINICAL TRIAL: NCT06513364
Title: A Phase Ib Randomized Parallel Study of Comparing WH002 With Paclitaxel Both Sequential of Epirubicin and Cyclophosphamide As Neoadjuvant Treatment of Women With HER2-Negative Breast Cancer
Brief Title: Neoadjuvant Chemotherapy With WH002 in Women With HER2-negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Wehand-Bio Pharmaceutical Co., Ltd (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WH002-I-102
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WH002 (Experimental): Group A（ddWH002-ddEC）：
  Regimen for Group A during Cycles 1-Cycles 4:
  • Paclitaxel Medium/Long-chain Fat Emulsion Injection (Cholesterol-Conjugated), 260 mg/m² administered intravenously on Day 1, with a cycle length of 2 weeks (Q2W), repeated for a total of 4 cycles.
  Regimen for Group A during Cycles 5-Cycles 8:
  • Epirubicin Hydrochloride 90 mg/m² and Cyclophosphamide for Injection 600 mg/m², both administered intravenously on Day 1, with each cycle lasting 2 weeks (Q2W), continued for 4 consecutive cycles.
  Interventions: Drug: WH002
- Paclitaxel Injection (Active Comparator): Group B (ddP-ddEC):
  Regimen for Group B during Cycles C1-C4:
  • Paclitaxel Injection (Paclitaxel®) 175 mg/m², administered intravenously on Day 1, with a cycle duration of 2 weeks (Q2W), repeated for a total of 4 cycles.
  Regimen for Group B during Cycles C5-C8:
  • Epirubicin Hydrochloride 90 mg/m² and Cyclophosphamide for Injection 600 mg/m², both administered intravenously on Day 1, with cycles recurring every 2 weeks (Q2W), for a series of 4 cycles.
  Interventions: Drug: paclitaxel injection

INTERVENTIONS:
Drug: WH002 — Group A（ddWH002-ddEC）： Regimen for Group A during Cycles 1-Cycles 4:WH002， 260 mg/m² administered intravenously on Day 1, with a cycle length of 2 weeks (Q2W), repeated for a total of 4 cycles.
  Regimen for Group A during Cycles 5-Cycles 8:
  • Epirubicin Hydrochloride 90 mg/m² and Cyclophosphamide for Injection 600 mg/m², both administered intravenously on Day 1, with each cycle lasting 2 weeks (Q2W), continued for 4 consecutive cycles.
  Other Names: Paclitaxel Medium/Long-chain Fat Emulsion Injection (Cholesterol-Conjugated)
  Arms: WH002
Drug: paclitaxel injection — Group B (ddP-ddEC):
  Regimen for Group B during Cycles C1-C4:
  • Paclitaxel Injection (Paclitaxel®) 175 mg/m², administered intravenously on Day 1, with a cycle duration of 2 weeks (Q2W), repeated for a total of 4 cycles.
  Regimen for Group B during Cycles C5-C8:
  • Epirubicin Hydrochloride 90 mg/m² and Cyclophosphamide for Injection 600 mg/m², both administered intravenously on Day 1, with cycles recurring every 2 weeks (Q2W), for a series of 4 cycles.
  Other Names: Taxol
  Arms: Paclitaxel Injection

SUMMARY:
The purpose of this study is to compare the safety and efficacy of bi-weekly WH002(Paclitaxel Medium and Long Chain Fat Emulsion Injection,Cholesterol Bound) vs Paclitaxel both followed by bi-weekly Epirubicin and Cyclophosphamide as neoadjuvant treatment in women with HER2-negative breast cancer.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open-label, positive-drug parallel-controlled phase Ib trial. The primary aim of this study was to compare the safety, efficacy, and pharmacokinetics of a dose-dense regimen of bi-weekly WH002 followed by bi-weekly epirubicin and cyclophosphamide (ddWH002-ddEC) versus bi-weekly Paclitaxel® followed by bi-weekly EC (ddP-ddEC) as neoadjuvant treatment in women with HER2-negative high-risk early-stage and locally advanced breast cancer. Patients randomly assigned to ddP-ddEC received premedication with oral prednisolone (12 and 6 hours before paclitaxel), IV dexchlorpheniramine, and cimetidine or ranitidine (30 minutes before paclitaxel). Whereas all of these premedication was not required in the ddWH002-ddEC group before receiving WH002.

Eligible subjects are those with biopsy-confirmed, HER2-negative breast cancer as verified by the research center, and whose tumor staging, as determined by imaging, falls into the categories of early high-risk (T1c-2, N1; T2, N0) or locally advanced (T1c-2, N2-3; T3-4, N0-3). Upon fulfilling all inclusion and exclusion criteria, participants will be randomized in a 1:1 ratio to either the WH002 followed by EC group (Group A) or the Paclitaxel® followed by EC group (Group B).Stratified randomization between the two groups based on tumor molecular subtypes:

* Luminal type (HER2-negative, ER or progesterone receptor positive),
* Triple-negative (HER2-negative, ER and progesterone receptor negative).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, female;
2. Histologically confirmed, untreated, unilateral primary invasive breast cancer;
3. Confirmed as HER2-negative breast cancer based on pathology testing at the research center; simultaneous determination of hormone receptor status (estrogen receptor [ER] and progesterone receptor [PgR]), tumor grade, and Ki67 value;
4. Clinical staging based on imaging assessment meeting any of the following criteria: IIA (T1c, N1; T2, N0), IIB (T2, N1; T3, N0), IIIA-IIIC (T1c-2, N2-3; T3, N1-3; T4, any N);
5. Patient agrees to undergo breast cancer surgery after completing neoadjuvant chemotherapy;
6. The Eastern Cooperative Oncology Group performance status ≤1;
7. Essentially normal function of major organs, with laboratory test values during screening conforming to the following standards:

   System Laboratory Test Values Hematology Absolute Neutrophil Count ≥1.5×10^9/L Platelets ≥100×10^9/L Hemoglobin ≥100g/L Kidney Serum Creatinine (Cr) ≤1.5×ULN or Creatinine Clearance (CCr) ≥60 mL/min (calculated using the Cockcroft-Gault formula) Liver Total Bilirubin (serum) ≤1.5×ULN Aspartate Aminotransferase and Alanine Aminotransferase ≤2.5×ULN Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5×ULN, unless the subject is on anticoagulant therapy；
8. Echocardiographic assessment: Left Ventricular Ejection Fraction (LVEF) ≥50%;
9. For patients of childbearing potential: Patients must agree to effective contraception during the treatment period and for at least 90 days after the last dose of study treatment, adopting double-barrier contraceptive methods, such as condoms, oral or injectable contraceptives, intrauterine devices, etc.;
10. Voluntarily signs the informed consent form, demonstrating good compliance.

Exclusion Criteria:

1. Patients with stage IV metastatic breast cancer or those deemed by the investigator as ineligible for curative surgical resection following neoadjuvant therapy;
2. Inflammatory breast cancer and bilateral primary breast cancer (including invasive and in situ carcinomas).
3. Patients requiring concurrent use of medications that may affect the metabolism of the study drug within 2 weeks prior to enrollment or during the study, such as strong CYP2C8 or CYP3A4 inducers or inhibitors;
4. Breast cancer patients who have previously received anti-tumor treatments, including radiotherapy, chemotherapy, endocrine therapy, targeted therapy, immunotherapy, or who have undergone breast surgery (excluding diagnostic biopsy for primary breast cancer);
5. Patients who must receive additional anti-tumor therapies other than the investigational product during the study, such as chemotherapy, endocrine therapy, targeted therapy, immunotherapy regimens, or radiotherapy;
6. Patients with a history of allergic constitution (excluding mild, asymptomatic seasonal allergies), or known hypersensitivity to taxane drugs/WH002 or its excipients [e.g., allergy to medications containing polyoxyethylated castor oil (like cyclosporine); or allergy to drugs containing hardened castor oil (such as vitamin injections); or allergy to lipid emulsion-based drugs], or known allergy to epirubicin, cyclophosphamide, and/or their excipients;
7. Patients with severe organ dysfunction (heart, lung, liver, kidney, brain, etc.), or those who have experienced severe cardiovascular events within 6 months prior to dosing, such as myocardial infarction, unstable angina, coronary artery bypass or peripheral arterial bypass graft surgery, congestive heart failure, significant cerebrovascular events (including transient ischemic attacks), or have arrhythmias requiring treatment, confirmed prolongation of QTc interval (≥470ms) upon reassessment, and chronic heart failure patients (NYHA class III and IV); poorly controlled diabetes (fasting blood glucose ≥13.3mmol/L); inadequately controlled hypertension (systolic pressure >160 mmHg or diastolic pressure >100 mmHg), etc.;
8. Patients who have had or concurrently have other malignant tumors within the past 5 years, excluding those with basal cell or squamous cell carcinoma of the skin treated with curative intent, or cervical carcinoma in situ;
9. Patients with active infections requiring intravenous antibiotic treatment;
10. Women of childbearing potential who are pregnant, breastfeeding, or have a positive pregnancy test;
11. History of motor or sensory neuropathy from any cause (greater than NCI-CTCAE V5.0 Grade 1) prior to enrollment;
12. Participation in another clinical trial within 4 weeks prior to enrollment;
13. Any condition, as judged by the investigator, that makes the subject unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
All reported adverse events, serious adverse events and the percentage of drug-related adverse events, serious adverse events during the treatment period. | From the first administration of the medication until 28 days after the breast cancer surgery, or 28 days after the last administration of the medication.
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported.Compare the safety and tolerability between the WH002 group and the Paclitaxel® group during the treatment period. Patients will be assessed for adverse events by clinical examination, questioning for symptoms of toxicity, laboratory assessments, vital signs, ECG and LVEF.
  Neurological toxicity and other toxicities will be assessed throughout the study according the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
pathologic Complete Response(pCR) Rate | the duration of 28 days of Postoperative of Breast Cancer；
  Comparison of the overall pathological complete response rate (tpCR, defined as ypT0/ypTis ypN0) between the WH002 group and the Paclitaxel® group;
pathologic Complete Response (pCR) and Breast Pathological Complete Response Rate(bpCR ) | the duration of 28 days of Postoperative Breast Cancer；
  Comparison of the rates of pCR defined as ypT0 ypN0 and bpCR (ypT0/Tis) between the WH002 group and the Paclitaxel® group;
objective response rate(ORR) | At the end of Cycle 2 (each cycle is 14 days)； At the end of Cycle 4 (each cycle is 14 days)；At the end of Cycle6 (each cycle is 14 days)；At the end of Cycle 8 (each cycle is 14 days)；
  Comparison of the objective response rate (ORR) assessed by ultrasound, mammography or MRI after paclitaxel treatment and sequential EC treatment between the WH002 group and the Paclitaxel® group;
time to peak concentration (Tmax) | the 1th day and 2th day of cycle 1 (each cycle is 14 days)，the 1th day and 2th day of cycle 4 (each cycle is 14 days)；
  Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.
peak concentration (Cmax) | cycle 1（14 days）and cycle 4（14 days）；
  Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.
AUC0-inf | cycle 1（14 days）and cycle 4（14 days）；
  area under the concentration-time curve from time zero to the infinity. Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.
AUC0-t | cycle 1（14 days）and cycle 4（14 days）；
  area under the concentration-time curve from time zero to the last measurable .Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.
half-life (t½) | cycle 1（14 days）and cycle 4（14 days）；
  Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.
clearance (CL) | cycle 1（14 days）and cycle 4（14 days）；
  Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.
free fraction | cycle 1（14 days）and cycle 4（14 days）；
  ratio of free paclitaxel concentration to total paclitaxel concentration. Comparison of pharmacokinetic parameters of total and unbound paclitaxel between the WH002 group and the Paclitaxel® group following drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, MD, Principal Investigator — National Cancer Center/Cancer Hospital, Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No